CLINICAL TRIAL: NCT00403780
Title: Pregabalin for Pain Reduction in Critical Limb Ischemia - A Double Blind, Randomized Controlled Study
Brief Title: Randomized Study of Pregabalin for Pain Reduction in Patients With Rest Pain and Lower Limb Ischemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low inclusion rate
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Jonas Malmstedt, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREPARED_00
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Critical Limb Ischemia; Arterial Occlusive Disease; Pain; Ischemia
Keywords: Critical limb ischemia; Pain control; Rest pain in lower limb ischemia; pregabalin; randomized controlled study; Ischemia, therapy; Lower extremity, blood supply; Pain, prevention & control; Pain, therapy
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Arterial Occlusive Diseases; Pain; Ischemia; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Active intervention with pregabalin
  Interventions: Drug: pregabalin
- B (Placebo Comparator): placebo arm with capsule Lyrica Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — Capsule pregabalin 75 mg once or twice daily up to a total dose of 600mg daily (300mg twice daily) for a total of minimum 14 days and maximum 8 weeks.
  Dosage will be up titrated during first study week according to a prespecified scheme, starting with one capsule daily.
  Other Names: Capsule Lyrica 75mg. Manufacturer company: Pfizer
  Arms: A
Drug: placebo — Capsule placebo once or twice daily up to a total dose of 8 capsules(4 capsules twice daily) for a total of minimum 14 days and maximum 8 weeks. Dosage will be up titrated during first study week according to a prespecified scheme, starting with one capsule daily.
  Other Names: Lyrica Placebo
  Arms: B

SUMMARY:
The hypothesis behind the trial is the concept that Pregabalin is effective in reducing pain at rest in lower limb ischemia, and the study evaluates active treatment or placebo added to the regular pain regimens for these patients.

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) is the end stage of peripheral arterial disease in the legs and is a consequence of deteriorating blood flow supply to the lower limbs. The clinical definition of CLI includes peripheral arterial disease and recurrent rest pain for at least two weeks with or without ulcers or gangrene.

In patients not amenable to revascularization - around 35% - amputation or palliative conservative care remains the options. Pain control is a vital part of any treatment of these patients. Besides being the principal conservative treatment, also patients undergoing revascularization experience severe pain both during work up and after surgery.

Experimental data indicate that pain in CLI is multimodal and to a large extent neuropathic. Still, current therapy is mostly based on opioid treatment, which clinically often affects pain moderately. The doses required to influence pain are also associated to severe side effects. Accordingly, there is a great need to improve pain control in the rather common disease CLI.

comparisons: pregabalin up to 600mg daily in addition to regular pain regimens compared to placebo and regular pain regimens.

ELIGIBILITY:
Inclusion Criteria:

* Rest pain, gangrene or ulcers located below the patella for a duration of at least two weeks (either one of these criteria are sufficient).
* One measurement of: Ankle blood pressure(ABP) <70 mm Hg, an toe blood pressure(TBP) <50, or a TcPO2<45 mm Hg, or an ankle/brachial pressure index <0.7 (either one of these criteria are sufficient).
* Informed consent obtained

Exclusion Criteria:

* Age < 55 years
* Women of childbearing potential
* Patients already medicating with Pregabalin or Gabapentin
* Creatinine clearance <30ml/min
* Amputation necessary within two weeks
* Revascularization necessary within two weeks (open vascular surgery or endovascular)
* A medical history of clear dizziness
* NYHA class IV heart failure
* Known hypotension, or having a systolic arm blood pressure <120 mm Hg (two consecutive measurements with the patient lying supine)
* Simultaneous or previous (within 30 days prior to study entry participation in a clinical study using experimental drugs or devices
* Mental condition making the subject unable to understand the concepts and risk of the study
* Known allergies against pregabalin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-06; Primary Completion 2013-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Reduction in Rating Scale (RS) pain compared to baseline. RS Pain will be assessed at 7, 14 days for all participants and after 28 and 56 days for patients continuing the extended phase of study. | 1, 2, 4 and 8 weeks after randomization

SECONDARY OUTCOMES:
Improvement in the Short Form 36 (SF-36) parameter "bodily pain". | This parameter will be evaluated at baseline, after seven and 14 days of treatment. Patients continuing in the study will be scored also at 28 and 56 days.
The amount, dose and duration of concomitant pain medication use during study compared to use before study. | 2 weeks after randomization
Safety outcomes and adverse events will be examined and recorded throughout the study. Patient reported dizziness will be recorded separately in the CRF, as well as blood pressure at visits. | up to 8 weeks, as long as patients is in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wahlberg, MD. PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Deptartment of Vascular Surgery, Sahlgrenska University Hospital, Gothenburg
  - Department of Vascular Surgery, Karolinska University Hospital, Stockholm
  - Deptartment of Surgery, South Hospital, Stockholm

REFERENCES:
- [Background] Caraceni A, Zecca E, Bonezzi C, Arcuri E, Yaya Tur R, Maltoni M, Visentin M, Gorni G, Martini C, Tirelli W, Barbieri M, De Conno F. Gabapentin for neuropathic cancer pain: a randomized controlled trial from the Gabapentin Cancer Pain Study Group. J Clin Oncol. 2004 Jul 15;22(14):2909-17. doi: 10.1200/JCO.2004.08.141. PMID 15254060
- [Background] Hultgren R, Olofsson P, Wahlberg E. Sex-related differences in outcome after vascular interventions for lower limb ischemia. J Vasc Surg. 2002 Mar;35(3):510-6. doi: 10.1067/mva.2002.120043. PMID 11877700